CLINICAL TRIAL: NCT05518942
Title: Effects of Sensorimotor Rhythm Neurofeedback on Insomnia in Patients With Benign Brain Tumors Underwent Surgery
Brief Title: Effects of SMR Neurofeedback on Insomnia in Patients With Benign Brain Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting cases due to the epidemic
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202200998B0A3
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Benign Brain Tumor; Neurofeedback; Insomnia
MeSH Terms: conditions — Brain Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensorimotor rhythm neurofeedback training (Experimental): Sensory motor rhythm neurofeedback: The subjects will perform 60 minutes per week for 10 weeks, with a total training time of 600 minutes. The intervention in this trial lasts for 10 weeks (1 time/week), with the goal of improving sensory motor rhythm. Since this training uses visual and auditory feedback, if patients are assigned to this group, they will be ask to wear an EEG cap with 19 electrodes. They can take a relaxed sitting posture and choose animations (e.g., puzzles, mazes, and other feedback content), and then focus on computer screen animation for training, each training time is approximately 60 minutes.
  Interventions: Behavioral: sensorimotor rhythm neurofeedback training
- control group (No Intervention): Patient should maintain their usual activity and treatment. Research assistants will weekly contact them to confirm their compliance.

INTERVENTIONS:
Behavioral: sensorimotor rhythm neurofeedback training — In this study, baseline brain waves will be recorded for 5 minutes before each treatment, and the average value of SMR waves was used as the basis for setting the treatment threshold for the week. During the treatment, the subjects are arranged to sit in front of a computer screen with a game or animation playing. The individual focuses on the games or animations on the screen. The software will analyze the brain wave signals from the brain and convert them into visual and auditory feedback on the computer screen. Clients can learn to control brain activity and give visual and auditory feedback when a set threshold is reached
  Arms: sensorimotor rhythm neurofeedback training

SUMMARY:
Insomnia is the most common sleep disorder in patients with primary brain tumors. In the past, 21.5% to 59.2% of patients with primary brain tumors suffer from insomnia symptoms. In addition to hypnotics, nonpharmacological interventions for insomnia in patients with brain tumors are still lacking. When using hypnotics may cause daytime sleepiness, cognitive impairment, and increase the risk of cancer, seeking an effective intervention is of clinical importance. Sensorimotor rhythm neurofeedback therapy has been shown to improve insomnia in different populations. However, its effect on insomnia has not been explored in patients with brain tumors. We, therefore, aim to investigate the feasibility and effect of sensorimotor rhythm neurofeedback in improving insomnia in patients with benign brain tumors after surgery and to examine the correlation between the degree of insomnia improvement and quality of life changes after receiving sensorimotor rhythm neurofeedback.

DETAILED DESCRIPTION:
Brain tumors are mainly divided into primary and metastatic, and are further divided into benign and malignant according to the pathological type. Among them, meningioma and pituitary tumor are the top two most common primary benign brain tumors, accounting for 36.1% respectively. -54.5% and 10-15%, while the most malignant glioblastoma accounts for 45-49.1% of primary malignant brain tumors. Among them, glioblastomas are more common in men and meningiomas are more common in women.

Insomnia is the most common sleep disorder in patients with primary brain tumors. Insomnia refers to difficulty falling asleep, staying awake and unable to fall asleep while sleeping, frequently waking up during sleep period or shortening sleep time, resulting in still feeling tired after getting up and affecting daily life functions. In the past, in terms of the prevalence of insomnia, primary brain 21.5%~59.2% of patients with tumor had insomnia symptoms, and if subdivided into benign, 46.8% of patients with primary benign brain tumor.

According to the results of the study, patients with primary brain tumors still have widespread and persistent insomnia problems after treatment, and even up to one year after surgery, there are still studies showing insomnia problems. Savard et al (2011) reported that insomnia is also a cancer A common and persistent problem among patients, the attack rate of insomnia generally decreased over time, but remained prevalent (36%) even at the end of 18 months. However, in real life, although insomnia has a high attack rate and a high burden on the family, and even affects the overall quality of life of patients, it is often not valued and treated.

Neurofeedback (NFB), also known as brain wave training, is a method to help subjects consciously control their brain waves. In order to reflect the state of brain activity, the software analyzes the measured brain waves and provides feedback signals to teach individuals to self-regulate brain waves. After repeated training, the target brain waves can be generated. When the threshold is reached, it will give visual and auditory feedback. Neurofeedback has been used clinically in many diseases and healthy individuals that cannot be effectively treated with drugs, such as insomnia, ADHD, epilepsy, fibromyalgia, depression, anxiety, pain, learning and memory, etc. For insomnia, the use of neurofeedback therapy can help people who usually take an hour or so to fall asleep fall asleep faster.

According to Lambert-Beaudet et al. (2021) reviewing the latest research on the use of neurofeedback in the treatment of insomnia, the enhancement of sensorimotor rhythm neurofeedback to improve insomnia was the most included and confirmed to improve insomnia. And multiple studies have confirmed that sensorimotor rhythm neurofeedback enhancement training can lead to increased sleep spindle density, decreased sleep onset latency, increased total sleep time, and decreased wake-up after falling asleep. Therefore, sensorimotor rhythm neurofeedback enhancement training can be an effective method for non-drug intervention in the treatment of insomnia. Given that the effects of sensorimotor rhythm neurofeedback training on insomnia have not been studied in patients with benign brain tumors after surgery, further studies in this group are warranted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as primary benign brain tumors such as: meningioma, schwannoma, pituitary tumor, craniopharyngioma according to the results of pathological tissue sections and has completed treatment such as : Surgery, radiation therapy, etc. for at least 7 days.
* Aged from 20 to 65 years old and conscious, able to communicate in Mandarin and Taiwanese.
* Cognitive ability sufficient to complete the questionnaire.
* Complaints of insomnia and ISI score ≥ 8

Exclusion Criteria:

* Long-term shift workers one month before the included study.
* Pregnant women.
* Jet lag workers, such as airline workers.
* Vision, hearing or motor dysfunction is severe enough to affect the participating researcher.
* Preoperative diagnosis of insomnia or long-term use of sleep aids or psychiatric drugs.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Changes in Insomnia Severity | at baseline and the 10th week after Intervention finished
  The ISI consists of seven items, and each item can be rated from 0 to 4, resulting in total score ranging from 0 to 28, with higher scores indicating greater insomnia severity. A cutoff score of > 7 is used to diagnose subthreshold insomnia.
Changes in Sleep parameters from sleep logs: sleep onset latency(SOL) | at baseline and the 10th week after Intervention finished
  Sleep onset latency(SOL) is the time of duration from lying on bed to fall asleep. SOL shorter than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: after sleep onset(WASO) | at baseline and the 10th week after Intervention finished
  Wake after sleep onset(WASO) is the total time of wakefulness after sleep onset. WASO less than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: total sleep time(TST) | at baseline and the 10th week after Intervention finished
  Total sleep time(TST) is the total time of falling asleep. TST will be used to calculate sleep efficiency(SE).
Changes in Sleep parameters from sleep logs: sleep efficiency(SE) | at baseline and the 10th week after Intervention finished
  Sleep efficiency(SE) is the percentage of total sleep time to time in bed. A good sleep condition should meet the criteria of SE greater than 85%.

SECONDARY OUTCOMES:
changes in quality of life | at baseline and the 10th week after Intervention finished
  The M.D. Anderson Syndrome Inventory-Taiwan Form (MDASI-Taiwan Form) is mainly used to assess the severity of various cancer symptoms in cancer patients due to cancer disease itself and various cancer treatments. The item, divided into two parts, the first part is the severity of cancer symptoms (symptom intensity): 0 points means no symptoms, 10 points means the most severe degree you can imagine, 1-3 points are mild, 4-6 points are mild Moderate, a score of 7 or more is severe; Part II: Severity of cancer symptoms that interfere with the functioning of life activities (life interference intensity): 0 means no interference, 10 means complete interference, and 1-3 means mild , 4 - 6 as moderate, 7 or more as severe.
Changes in Depression | at baseline and the 10th week after Intervention finished
  Depression will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of depression. The total score should be multiplied by 2 range from 0-42, if score>9 is associated with depression. The higher score means more severe depression
Changes in Anxiety | at baseline and the 10th week after Intervention finished
  Anxiety will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of anxiety. The total score should be multiplied by 2 range from 0-42, if score>7 is associated with anxiety. The higher score means more severe anxiety.
Changes in Stress | at baseline and the 10th week after Intervention finished
  Stress will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of stress. The total score should be multiplied by 2 range from 0-42, if score>14 is associated with anxiety. The higher score means more severe stress

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital., Taipei, Taiwan